CLINICAL TRIAL: NCT03819205
Title: Investıgatıng the Effect of Kinesiotaping on Hand Functions in Children With Cerebral Palsy
Brief Title: Is Kinesio Taping Treatment Effective in Children With Cerebral Palsy?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, ZEYNEP TOKEL, : Principal investigator, Dokuz Eylul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DorkuzEUZTOKEL
Record Dates: First submitted 2019-01-23; First posted 2019-01-28 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; upper extremity kinesiotaping; modified house
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: self-controlled study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- kinesiotaping group(before/after) (Experimental): * Hemiplegic CP:Kinesiotaping on the affected side
  * Diplegic, tetraplegic CP: side of upper extremity which children have been used to but have obstacles in daily life
  * intervention Duration: For 1 week at least 2-3 hours a day, renewing if it's necessary.
  * Note:Patients will be also recomended dealing with the grasping and releasing activities in daily living at about 2-3 hours a day.
  * Evaluation: In a way that every patient has to be the control of themselves, 1 week before kinesiotaping, immediately after kinesiotaping and 1 week after the period of kinesiotaping, patients will be evaluated with box and block test, nine hole peg test, modified house clasification and the active/passive wrist dorsiflexion range of motion
  Interventions: Other: kinesiotaping

INTERVENTIONS:
Other: kinesiotaping — The participants will receive kinesiotaping treatment on the affected side for the hemiplegic CP's and for diplegic, tetraplegic CP's the side of upper extremity which children have been used to but have obstacles in daily life for 1 week at least 2-3 hours a day, renewing if it's necessary. The participants will be also recomended dealing with the grasping and releasing activities in daily living at about 2-3 hours a day. In a way that every patient has to be the control of themselves, 1 week before kinesiotaping, immediately after kinesiotaping and 1 week after the period of kinesiotaping, patients will be evaluated with box and block test, nine hole peg test, modified house clasification and the active/passive wrist dorsiflexion range of motion

SUMMARY:
Cerebral palsy (CP) is defined as a non-progressive lesion of the immature brain. Children with CP may present with a variety of motor impairments.

The impaired upper limb function of children with cerebral palsy (CP) limits and restricts participation in activities of daily living.

Kinesio Taping (KT) is commonly used in sport injuries, in neurology and oncology patients following the surgical protocols, and for pediatric rehabilitation to reduce pain, facilitate or inhibit muscle activity, prevent injuries, reposition joints, aid the lymphatic system, support postural alignment, and improve proprioception. Kinesiotaping is a treatment that has not been studied much and can be applied in cerebral palsy. The tapes were grouped as elastic and rigid. In fact, there has been a few studies that investigates the effect of upper extremity elastic kinesiotaping. High methodological studies about its efficacy in this population are rare.

DETAILED DESCRIPTION:
34 Children with cerebral palsy aged between 6-18 applied to Dokuz Eylül Üniversity Medical School Hospital Physical Medicine ve Rehabilitation Department will be included the study. Patients have diagnosed as CP with the subgroup of diplegic, hemiplegic, tetraplegic and mixt. The upper extremity side will be chosen as the affected side for the hemiplegic CP's and for diplegic, tetraplegic CP's the side of upper extremity which children have been used to but have obstacles in daily life. The chosen upper extremity side will be taped with the functional correction technique on the dorsum of the hand and forearm by clinician. Patients will be taped at least 2-3 hours a day every day and they will be also recomended dealing with the grasping and releasing activities in daily living at about 2-3 hours a day. In a way that every patient has to be the control of themselves, 1 week before kinesiotaping, immediately after kinesiotaping and 1 week after the period of kinesiotaping patients will be evaluated with box and block test, nine hole peg test, modified house clasification score and the active/passive wrist dorsiflexion range of motion. The investigator will also note the gross motor function clasification system level, dominant hand side and affected side, for chosen upper extremity side's zancolli clasification, modified aschwort scale of wrist and hand fingers, manual ability clasification system level for every patient.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 6-18
2. Following up with diagnose of hemiplegic/diplegic/tetraplegic CP patients with current imaginig findings
3. Patient with stable clinical status
4. Stage ≤2 patients depended on the modified ascwort scale
5. Patients who are eligible to participate the study tests with suitable cognitive state
6. Patients who agreed to participate the study.

Exclusion Criteria:

1. Stage >2 patients depended on the modified ascwort scale
2. Botilinum toxin intervention to the upper extremity in the last 6 months.
3. Patients who undergo upper extremity surgery.
4. Patients who have contraindication for kinesiotaping (Wide and severe skin injury, open wounds at risk of infection , allergic reactions)
5. Patients with intense sensory and motor loss in the banding area
6. Patients classified in stage IIB and above according to Zancolli stage

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Estimated)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-03-10 (Estimated); Study Completion 2019-03-10 (Estimated)

PRIMARY OUTCOMES:
Box and block test | 1 week before kinesiotaping and 1 week after the period of kinesiotaping (change form baseline will be evaluated)
  With the stopwatch, it is recorded how many small cubes are transferred to the other side of the box within 60 seconds.
Nine hole peg test | 1 week before kinesiotaping and 1 week after the period of kinesiotaping (change form baseline will be evaluated)
  A wooden box with nine holes is placed in front of the patient and held in seconds with the stopwatch. Insersion and extraction time of pegs in second are noted.

SECONDARY OUTCOMES:
Modified house clasification score | 1 week before kinesiotaping and 1 week after the period of kinesiotaping (change form baseline will be evaluated)
  The score obtained from the Modified House Classification is calculated by recording the patient's capabilities among the listed 32 activities
Active/passive wrist dorsiflexion range of motion | 1 week before kinesiotaping and 1 week after the period of kinesiotaping (change form baseline will be evaluated)
  With goniometer active/passive wrist dorsiflexion range of motion will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Tokel, MD, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, İ̇zmi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No